CLINICAL TRIAL: NCT04922970
Title: Strength Training as Prevention and Treatment of Late Effects in Long-term Survivors of Pediatric HSCT.
Acronym: STEPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other); Danish Child Cancer Foundation (Other); University of Copenhagen (Other); The Danish Cancer Research Foundation (Unknown)
Responsible Party: Principal Investigator, Klaus Gottlob Müller, Professor, Senior consultant, Doctor of Medical Science and ph.d., Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STEPS
Record Dates: First submitted 2021-06-04; First posted 2021-06-11 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Stem Cell Transplant; Late Effect; Metabolic Syndrome; Cardiovascular Diseases
Keywords: Strength training; Resistance training
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The same interventon will be applied to two groups, a group of previously recipients of bone marrow transplantation, and a group of age- and sex-matched controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Strength training (Experimental): In this arm participants will go through the "Strength training intervention".
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Strength training — The interventon consist of 3 weekly, supervised group sessions for 4 months (16 weeks). The sessions consist of progressive full body strength training with a primary focus on lower extremity muscle strength. The leg exercises are leg press, knee extension and leg curl. In addition, participants will perform two upper body exercises. Physical assessment will take place immediately and monthly until 4 months.

SUMMARY:
Today the overall survival of childhood cancers has increased to above 85%. This increase is partially caused by treatment with bone marrow transplantation. A bone marrow transplantation is an efficient treatment against high-risk leukemia, as well as other life-threatening immunological and hematological diseases. However, it is unfortunately also related to the risk of developing a long series of late effects during early adulthood, such as low muscle mass, cardiovascular disease and diabetes. Conditions known from the older generations of the general population and also conditions highly related to lifestyle factors in the general population.

In the group of survivors after bone marrow transplantation, the cause for these late effects is not fully understood, as the same close association to lifestyle factors as seen in the general population, is not present in this group. Multiple studies have examined the possible causes, and it have been shown that certain elements of a bone marrow transplantation, ie. total body irradiation, are associated with the risk of developing late effects. As the cause is not fully understood, it is not known whether the treatment and preventive strategies, that would be applied in the general population for these conditions, are effective in this group.

Therefore, in this study the investigators aim at examining the effect of a strength training intervention on the development of the aforementioned late effects to treatment with bone marrow transplantation during childhood.

The investigators will invite a group of persons, transplanted during childhood, as well as an age- and sex-matched control group to participate in the study. Both groups will go through a 16-week strength training intervention, and a thorough health examination before and after the intervention, to assess metabolic status and body composition.

If the investigators find a positive effect of strength training on muscle mass and risk factors for developing cardiovascular disease and diabetes in persons, treated with bone marrow transplantation during childhood, it will support the implementation of structured training programs in the follow-up of these patients. Thereby hopefully contributing to an increased quality of life, as well as an increased life expectancy in the group of survivors after bone marrow transplantation during childhood.

ELIGIBILITY:
Inclusion Criteria:

* Living in Copenhagen, Denmark or surrounding area - making it possible to engage in strength training 3 times a week at Bispebjerg Hospital, Copenhagen, Denmark.
* ≥ 18 years old

Exclusion Criteria:

* Illness or physical handicap making it impossible to participate in the training intervention
* Pregnancy
* Not Danish or English speaking
* Anemia
* Already performing regular structured physical training
* Strict vegan or vegetarian diet
* Illness or ongoing treatment that hinders study examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Changes in cross sectional area of m. quadricpes femoris. | 1 week pre intervention
  Muscle mass as measured by cross sectional area of m. quadriceps femoris at midthigh level, on an MRI scan.
Changes in cross sectional area of m. quadricpes femoris. | 1 week post intervention
  Muscle mass as measured by cross sectional area of m. quadriceps femoris at midthigh level, on an MRI scan.

SECONDARY OUTCOMES:
Changes in components of the Metabolic Syndrome: Waist circumference | 1 week pre intervention
  Waist circumference will be measured at the level of the superior border of the iliac crest, at the end of a normal expiration with a tape measure to the nearest 0.1 cm, as suggested by The US National Cholesterol Education Programme. Patients will be classified according to The US National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III) definition of the Metabolic Syndrome. We will report changes in the number of components fulfilled.
Changes in components of the Metabolic Syndrome: Waist circumference | 1 week post intervention
  Waist circumference will be measured at the level of the superior border of the iliac crest, at the end of a normal expiration with a tape measure to the nearest 0.1 cm, as suggested by The US National Cholesterol Education Programme. Patients will be classified according to The US National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III) definition of the Metabolic Syndrome. We will report changes in the number of components fulfilled.
Changes in components of the Metabolic Syndrome: Triglycerides | 1 week pre intervention
  Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand. Patients will be classified according to The US National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III) definition of the Metabolic Syndrome. We will report changes in the number of components fulfilled.
Changes in components of the Metabolic Syndrome: Triglycerides | 1 week post intervention
  Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand. Patients will be classified according to The US National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III) definition of the Metabolic Syndrome. We will report changes in the number of components fulfilled.
Changes in components of the Metabolic Syndrome: HDL-cholesterol | 1 week pre intervention
  Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand. Patients will be classified according to The US National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III) definition of the Metabolic Syndrome. We will report changes in the number of components fulfilled.
Changes in components of the Metabolic Syndrome: HDL-cholesterol | 1 week post intervention
  Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand. Patients will be classified according to The US National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III) definition of the Metabolic Syndrome. We will report changes in the number of components fulfilled.
Changes in components of the Metabolic Syndrome: Fasting glucose | 1 week pre intervention
  Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand. Patients will be classified according to The US National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III) definition of the Metabolic Syndrome. We will report changes in the number of components fulfilled.
Changes in components of the Metabolic Syndrome: Fasting glucose | 1 week post intervention
  Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand. Patients will be classified according to The US National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III) definition of the Metabolic Syndrome. We will report changes in the number of components fulfilled.
Changes in components of the Metabolic Syndrome: Blood pressure | 1 week pre intervention
  Blood pressure will be measured on the upper arm while sitting in the suppine position, after 10 minutes of rest, with an automated blood pressure monitor. Blood pressure will be measured three times, or untill there is less than 10 mmHg difference between measurements. The final blood pressure will be a mean of the two last measurements.
  Patients will be classified according to The US National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III) definition of the Metabolic Syndrome. We will report changes in the number of components fulfilled.
Changes in components of the Metabolic Syndrome: Blood pressure | 1 week post intervention
  Blood pressure will be measured on the upper arm while sitting in the suppine position, after 10 minutes of rest, with an automated blood pressure monitor. Blood pressure will be measured three times, or untill there is less than 10 mmHg difference between measurements. The final blood pressure will be a mean of the two last measurements.
  Patients will be classified according to The US National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III) definition of the Metabolic Syndrome. We will report changes in the number of components fulfilled.
Hip circumference | 1 week pre intervention
  Measurement of hip circumference at the widest part of the buttocks with a tape measure, to the nearest 0.1 cm.
Hip circumference | 1 week post intervention
  Measurement of hip circumference at the widest part of the buttocks with a tape measure, to the nearest 0.1 cm.
Urine sample - microalbuminurea | 1 week pre intervention
  A urine sample for analyses of microalbuminurea in mg/L.
Urine sample - microalbuminurea | 1 week post intervention
  A urine sample for analyses of microalbuminurea in mg/L.
Muscle strength of quadriceps femoris | 1 week pre intervention
  Rate of force development, maximal isometric and dynamic force capacity measured by KinCom Dynamometer
Muscle strength of quadriceps femoris | 1 week post intervention
  Rate of force development, maximal isometric and dynamic force capacity measured by KinCom Dynamometer
Handgrip strength | 1 week pre intervention
  Handgrip strength measured with handheld Dynamometer
Handgrip strength | 1 week post intervention
  Handgrip strength measured with handheld Dynamometer
Muscle performance: Timed-up-and-go | 1 week pre intervention
  Timed-up-and-go test: The participant sits on a chair, that allow the participant to flex the leg at a 90 degree angle, with the back against the chair and arms on the knees. From this position the participant stands up straight and walk 3 m, turns around and go back to the chair and sit down as fast as possible, time in seconds is the outcome. The lowest score of three consecutive tries will be used in the analysis.
Muscle performance: Timed-up-and-go | 1 week post intervention
  Timed-up-and-go test: The participant sits on a chair, that allow the participant to flex the leg at a 90 degree angle, with the back against the chair and arms on the knees. From this position the participant stands up straight and walk 3 m, turns around and go back to the chair and sit down as fast as possible, time in seconds is the outcome. The lowest score of three consecutive tries will be used in the analysis.
Muscle performance: Sit-to-stand 30 sec. | 1 week pre intervention
  Sit-to-Stand 30 sec: The participant sits on a chair allowing the participant to flex the legs at a 90 degree angle. The participant is instructed to stand up straight, and return to sitting, as many times as possible in 30 sec. The arms should be crossed in front of the body or hanging by the side. Number of repititions is the outcome.
Muscle performance: Sit-to-stand 30 sec. | 1 week post intervention
  Sit-to-Stand 30 sec: The participant sits on a chair allowing the participant to flex the legs at a 90 degree angle. The participant is instructed to stand up straight, and return to sitting, as many times as possible in 30 sec. The arms should be crossed in front of the body or hanging by the side. Number of repititions is the outcome.
Muscle performance: Sit-to-stand 60 sec. | 1 week pre intervention
  Sit-to-Stand 60 sec: The participant sits on a chair allowing the participant to flex the legs at a 90 degree angle. The participant is instructed to stand up straight, and return to sitting, as many times as possible in 60 sec. The arms should be crossed in front of the body or hanging by the side. Number of repititions is the outcome.
Muscle performance: Sit-to-stand 60 sec. | 1 week post intervention
  Sit-to-Stand 60 sec: The participant sits on a chair allowing the participant to flex the legs at a 90 degree angle. The participant is instructed to stand up straight, and return to sitting, as many times as possible in 60 sec. The arms should be crossed in front of the body or hanging by the side. Number of repititions is the outcome.
Cardiorespiratory fitness: 6 minute walk test | 1 week pre intervention
  6 min. walk test: The participant walks as far as possible on a 15 m lane in 6 min. Distance in meters is the outcome.
Cardiorespiratory fitness: 6 minute walk test | 1 week post intervention
  6 min. walk test: The participant walks as far as possible on a 15 m lane in 6 min. Distance in meters is the outcome.

OTHER OUTCOMES:
Histology of thigh muscle | 1 week pre intervention
  Muscle biopsy sampled from the vastus lateralis muscle, with a Bergstroem needle with manual suction.
Histology of thigh muscle | 1 week post intervention
  Muscle biopsy sampled from the vastus lateralis muscle, with a Bergstroem needle with manual suction.
Body composition: Intraabdominal visceral fat | 1 week pre intervention
  Amount of visceral fat intraabdominally, as measured on a multisectional MRI scan from diaphragma to the pelvis with Dixon sequences.
Body composition: Intraabdominal visceral fat | 1 week post intervention
  Amount of visceral fat intraabdominally, as measured on a multisectional MRI scan from diaphragma to the pelvis with Dixon sequences.
Body composition: Abdominal subcutaneous fat | 1 week pre intervention
  Amount of subcutaneous fat in the abomen region, as measured on a multisectional MRI scan from diaphragma to the pelvis with Dixon sequences.
Body composition: Abdominal subcutaneous fat | 1 week post intervention
  Amount of subcutaneous fat in the abomen region, as measured on a multisectional MRI scan from diaphragma to the pelvis with Dixon sequences.
Body composition: Hepatic fat | 1 week pre intervention
  Amount of hepatic fat (%), as measured on a MRI scan fromof the liver with Dixon sequences.
Body composition: Hepatic fat | 1 week post intervention
  Amount of hepatic fat (%), as measured on a MRI scan fromof the liver with Dixon sequences.
Body composition: Fat mass | 1 week pre intervention
  Body fat mass (%) will be analyzed on a whole-body DEXA scan
Body composition: Fat mass | 1 week post intervention
  Body fat mass (%) will be analyzed on a whole-body DEXA scan
Body composition: Fat free mass | 1 week pre intervention
  Fat free mass (%), as a surrogate measure of lean mass, will be analyzed on a whole-body DEXA scan
Body composition: Fat free mass | 1 week post intervention
  Fat free mass (%), as a surrogate measure of lean mass, will be analyzed on a whole-body DEXA scan
Body composition: Android-gynoid ratio | 1 week pre intervention
  Android-gynoid ratio will be calculated, as a ratio of the fat mass in the abdominal region and the fat mass in the hip area, obtained by a whole-body DEXA scan
Body composition: Android-gynoid ratio | 1 week post-intervention
  Android-gynoid ratio will be calculated, as a ratio of the fat mass in the abdominal region and the fat mass in the hip area, obtained by a whole-body DEXA scan
Body composition: Bone mineral density | 1 week pre intervention
  Bone mineral density, will be analyzed on a whole-body DEXA scan. Z- and T-scores will be calculated.
Body composition: Bone mineral density | 1 week post intervention
  Bone mineral density, will be analyzed on a whole-body DEXA scan. Z- and T-scores will be calculated.
Body mass index (BMI) | 1 week pre intervention
  BMI will be calculated based on measurements of height and weight. To measure height the participants will stand up straight against a wall, in bare feet looking straight forward, and will be measured to the nearest 0.1 cm. Weight will be measured on an automated weight wearing only light indoor clothing with empty pockets and no shoes. BMI is calculated as wieght in kg diveded by height in meters squared.
Body mass index (BMI) | 1 week post intervention
  BMI will be calculated based on measurements of height and weight. To measure height the participants will stand up straight against a wall, in bare feet looking straight forward, and will be measured to the nearest 0.1 cm. Weight will be measured on an automated weight wearing only light indoor clothing with empty pockets and no shoes. BMI is calculated as wieght in kg diveded by height in meters squared.
Total-cholesterol | 1 week pre intervention
  Will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Total-cholesterol | 1 week post intervention
  Will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
LDL-cholesterol | 1 week pre intervention
  Will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
LDL-cholesterol | 1 week post intervention
  Will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Adipokines: Adiponectin | 1 week pre intervention
  Will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Adipokines: Adiponectin | 1 week post intervention
  Will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Adipokines: Leptin | 1 week pre intervention
  Will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Adipokines: Leptin | 1 week post intervention
  Will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Growth factors | 1 week pre intervention
  Growth factors, i.e. IGF-1 and IGFBP-3, will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Growth factors | 1 week post intervention
  Growth factors, i.e. IGF-1 and IGFBP-3, will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Thyroid hormones | 1 week pre intervention
  Thyroid hormones, free triiodothyronine (T3) and thyroxine (T4) as well as thyroid stimulating hormone (TSH) will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Thyroid hormones | 1 week post intervention
  Thyroid hormones, triiodothyronine (T3) and thyroxine (T4) as well as thyroid stimulating hormone (TSH) will be analyzed in a plasma sample. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Sex hormones | 1 week pre intervention
  Analyses of sex hormones, including testosterone and estrogen levels. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Sex hormones | 1 week post intervention
  Analyses of sex hormones, including testosterone and estrogen levels. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Markers of inflammation | 1 week pre intervention
  Analyses of markers of inflammation, including high sensitivity CRP and IL-6 levels. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Markers of inflammation | 1 week post intervention
  Analyses of markers of inflammation, including high sensitivity CRP and IL-6 levels. Blood samples will be drawn from a cannual placed in an antecubital vein or a dorsal vein in the hand.
Oral glucose tolerance test: Glucose | 1 week pre intervention
  Analyses of plasma glucose levels during a 3 hour oral glucose tolerance test. Blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Glucose | 1 week post intervention
  Analyses of plasma glucose levels during a 3 hour oral glucose tolerance test. Blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Insulin | 1 week pre intervention
  Analyses of plasma insulin levels during a 3 hour oral glucose tolerance test. Blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Insulin | 1 week post intervention
  Analyses of plasma insulin levels during a 3 hour oral glucose tolerance test. Blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: C-peptide | 1 week pre intervention
  Analyses of plasma insulin levels during a 3 hour oral glucose tolerance test. Blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: C-peptide | 1 week post intervention
  Analyses of plasma insulin levels during a 3 hour oral glucose tolerance test. Blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Gut hormones | 1 week pre intervention
  Analyses of plasma levels of gut hormones, including GLP-1, GIP and glucagon during a 3 hour oral glucose tolerance test. Blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Gut hormones | 1 week post intervention
  Analyses of plasma levels of gut hormones, including GLP-1, GIP and glucagon during a 3 hour oral glucose tolerance test. Blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Bone remodeling markers | 1 week pre intervention
  Analyses of plasma levels of bone remodeling markers, including CTX and P1NP during a 3 hour oral glucose tolerance test. Blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Bone remodeling markers | 1 week post intervention
  Analyses of plasma levels of bone remodeling markers, including CTX and P1NP during a 3 hour oral glucose tolerance test. Blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Health related quality of life - SF36 | 1 week pre intervention
  Measure of health related quality of life, by the validated questionnaire SF-36. Outcome will be total score based o the questionnaire.
Health related quality of life - SF36 | 1 week post intervention
  Measure of health related quality of life, by the validated questionnaire SF-36. Outcome will be total score based o the questionnaire.
Accelerometry using actigraph | 1 week pre intervention
  measure of physical activity and sedentary behavior measured over 7 days recorded as counts per day
Accelerometry using actigraph | 1 week post intervention
  measure of physical activity and sedentary behavior measured over 7 days recorded as counts per day and minutes in moderate to vigorous activity
Oral glucose tolerance test: Matsuda Index | 1 week pre intervention
  Based on glucose and insulin values from the OGTT the Matsuda Index will be calculated, as a measure of peripheral insulin sensitivity. For the OGTT blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Matsuda Index | 1 week post intervention
  Based on glucose and insulin values from the OGTT the Matsuda Index will be calculated, as a measure of peripheral insulin sensitivity. For the OGTT blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Insulinogenic Index | 1 week pre intervention
  Based on glucose and insulin values from the OGTT the insulinogenic Index will be calculated, as a measure of beta-cell function. For the OGTT blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Insulinogenic Index | 1 week post intervention
  Based on glucose and insulin values from the OGTT the insulinogenic Index will be calculated, as a measure of beta-cell function. For the OGTT blood samples will be drawn before and 7, 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the intake of 75 g of glucose disolved in 250 ml of water.

REFERENCES:
- [Derived] Krogh LM, Nissen A, Weischendorff S, Hartmann B, Andersen JL, Holst JJ, Sorensen K, Fridh MK, Mackey AL, Muller K. Bone remodeling in survivors of pediatric hematopoietic stem cell transplantation: Impact of heavy resistance training. Pediatr Blood Cancer. 2024 Sep;71(9):e31159. doi: 10.1002/pbc.31159. Epub 2024 Jul 2. PMID 38953152